CLINICAL TRIAL: NCT01038219
Title: Reliability of Subjective Assessment of Fever by Parents and Health Care Providers in Children and Adolescents
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC129-09CTIL
Record Dates: First submitted 2009-12-20; First posted 2009-12-23 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2014-05

CONDITIONS: FEVER
Keywords: fever; children; SUBJECTIVE ASSESSMENT
MeSH Terms: conditions — Fever

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- fever measurements: 1000 estimates and measurements of children's body temperatures will be carried out by parents and nurses in children's emergency and pediatric units as part of the routine work. The estimates and the measurements will be carried out on children who are referred to an emergency unit and who are hospitalized in the pediatric department-- both boys and girls of all ages. A patient might be measured several times.
  The measurements will be gathered in the course of one year. Before the routine taking of temperature, the accompanying parent will be asked to estimate the patient's temperature by feeling his forehead (with the back of the hand, the palm, lips). The parent will record his evaluation (without telling the nurse). Afterwards the nurse will do a similar evaluation (excepting the lip test), record it, and then the routine temperature measurement will be taken.

SUMMARY:
Background: Fever is a widespread symptom in many diseases. Therefore, its value and diagnostic importance are well known. Fever in children is one of the common reasons for a visit to the pediatrician. Also, taking temperature is a very simple action and accessible to the general public.

Temperature is measured in various parts of the body by using medical equipment. The type of method and thermometer varies according to the patient's age but often temperature is estimated by touch. Temperature measurement serves as a means for monitoring the patient's condition. For that reason, supervision of the body temperature is an important factor in the process of taking medical decisions.

Study rationale: the parent is often asked if the child's temperature has been taken. The most frequent answer is: "I didn't measure, but I felt that he has a temperature". The few studies carried out on this subject showed that many parents used touch to evaluate the child's body temperature, especially in infants.

Some studies checked the reliability of parents to estimate the child's body temperature by touch only. To the best of our knowledge, the reliability of medical staff (nurses) to estimate the child's body temperature by touch has never been studied.

The aim of the current study is to investigate whether parents and nurses correctly estimate the child's body temperature by touch, as compared to thermometer measurement during the pediatric unit's routine work.

DETAILED DESCRIPTION:
1000 estimates and measurements of children's body temperatures will be carried out by parents and nurses in the pediatric emergency unit and pediatric department as part of the routine work. The estimates and the measurements will be carried out on both boys and girls of all ages. A patient might be measured several times.

The measurements will be gathered in the course of one year. Before the routine taking of temperature, the accompanying parent will be asked to estimate the patient's temperature by feeling his forehead (with the back of the hand, the palm, lips). The parent will record his evaluation (without telling the nurse). Afterwards the nurse will perform a similar evaluation (excluding the lip test), record it, and then the routine temperature measurement will be taken and recorded.

Medical Equipment The temperature will be taken with the existing equipment in the emergency ward and in the children's ward. A rectal measurement will be taken in the case of children under two years old. Children over two will be measured orally. The temperature of children suffering from diarrhea and vomiting will be taken with an ordinary mercury thermometer. All other measurements will be made using an electronic, mobile thermometer manufactured by the Filac Company, (FasTemp electronic thermometer) routinely used in the emergency ward and pediatric departments.

ELIGIBILITY:
Inclusion Criteria:

* The estimates and the measurements will be carried out on children who are referred to an emergency unit and who are hospitalized in the pediatric department-- both boys and girls of all ages. A patient might be measured several times.

Exclusion Criteria:

* None

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children ages 0-18 years
  Boys and girls
Sampling Method: Non-Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2010-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
subjective assessment of fever by both parents and medical personnel will be unreliable | one year

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Meir MC, Kfar Saba
  - Pediatrics unit, Meir Medical Center, Kfar Saba